CLINICAL TRIAL: NCT06460415
Title: Effects of Photobiomodulation on Pain and Sexual Function in Women With Dyspareunia: Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Mariana Della Valentina Pessoa, Mariana Della Valentina Pessoa, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6.443.426
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Dyspareunia; Pain; Sexual Dysfunction
Keywords: photobiomodulation; dyspareunia; sexual dysfunction; physiotherapy; pelvic pain
MeSH Terms: conditions — Dyspareunia; Pain; Sexual Dysfunction, Physiological; Pelvic Pain

STUDY DESIGN:
Intervention Model Description: GPBM group - will receive application in 8 points (4 red and 4 infrared) in the vulvar region and 8 points (4 red and 4 infrared) in the intravaginal pelvic floor region of PBM and will be evaluated in the pre-intervention, post-intervention and in follow-ups of 15, 30, 90 and 180 days
  GS group - will receive simulation of PBM application in the same number of vulvar and intravaginal points, in the same places where it was applied in the GPBM group. and will be evaluated pre-intervention, post-intervention and in follow-ups of 15, 30, 90 and 180 days
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To control possible measurement biases in the present study, the following measures will be taken: all treatment sessions will be administered by the same trained and experienced researcher, to ensure that the treatment is homogeneous among the volunteers. The evaluators who will apply the scales, scores and questionnaires will be blinded to the allocation of volunteers to the groups under study. The sealed envelope method will be used for confidential allocation. Each envelope containing the allocated treatment will be sealed and numbered sequentially.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation group (GPBM) (Experimental): The volunteers in the GFBM group will undergo 8 sessions of a combined red and infrared laser protocol with 4J of infrared power and 4J of red power. Being applied at 8 points (4 red and 4 infrared) in the vulvar region and 8 points (4 red and 4 infrared) points in the intravaginal pelvic floor region.
  Interventions: Device: photobiomidulação
- Shan group (GS) (Placebo Comparator): The placebo control will be administered using the same device as the GFBM, but without any therapeutic dose delivery. Furthermore, the irradiated sites and irradiation time will be the same as PBMT. Volunteers will receive a total dose of 0 J in placebo mode. This treatment was also carried out in 8 sessions.
  For volunteers in the control group. There will be the possibility of them receiving treatment later if it proves effective in reducing pain.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: photobiomidulação — The volunteers in the GFBM group will undergo 8 sessions of a combined red and infrared laser protocol with 4J of infrared power and 4J of red power. Being applied at 8 points (4 red and 4 infrared) in the vulvar region and 8 points (4 red and 4 infrared) points in the intravaginal pelvic floor region. The MMO semiconductor laser device (GaA1As and InGaAlP) will be used with an area of the output laser beam at the NOZZLE of the laser pen of 3mm2 and wavelengths of 660nm (Red Laser) and 808nm (Infrared Laser) with a power of 100mW. The application will be carried out with the volunteers on a stretcher, in the supine position, gynecological position, with the knees and hips flexed and in abduction, feet supported on the stretcher.
  Arms: Photobiomodulation group (GPBM)
Other: Placebo — The placebo control will be administered using the same device as the GFBM, but without any therapeutic dose delivery. Furthermore, the irradiated sites and irradiation time will be the same as PBMT. Volunteers will receive a total dose of 0 J in placebo mode. This treatment was also carried out in 8 sessions.
  Arms: Shan group (GS)

SUMMARY:
The goal of this clinical trial is to compare the effects of vulvar and intravaginal application of PBM compared to the sham group on pain and sexual function in women with dyspareunia . The main question [s] it aims to answer are:

* What are the effects of vulvar and intravaginal application of photobiomodulation (PBM) compared to the sham group on the sexual function of women with dyspareunia in the immediate post-intervention moments and in follow-ups of 15, 30, 90 and 180 days?
* What are the effects of vulvar and intravaginal application of photobiomodulation (PBM) compared to the sham group on pain in women with dyspareunia in the immediate post-intervention moments and in follow-ups of 15, 30, 90 and 180 days?

Participants will The GPBM photobiomodulation group will receive, during the 8 days of intervention, application in 8 points (4 red and 4 infrared) in the vulvar region and 8 points (4 red and 4 infrared) in the intravaginal pelvic floor region of PBM while the GS group will receive simulation application of PBM in the same number of vulvar and intravaginal points, in the same places where it was applied in the GPBM group. To see if 8 applications of photobiomodulation are really capable of reducing pain and improving sexual function in women with dyspareunia

DETAILED DESCRIPTION:
Female sexual dysfunction is known as the disorder experienced by a woman when changes occur in her usual sexual behavior. It is estimated that between 16 and 40% of women suffer from some form of sexual dysfunction, and this percentage increases with age.1 Among the painful disorders, dyspareunia stands out, which is defined as pain perceived in the pelvis associated with sex with penetration. It can be applied to women and men. It usually occurs with penile penetration, but is often associated with pain during the insertion of any object. It can apply to anal and vaginal intercourse. It is classically subdivided into superficial, when it affects the vulva and vaginal entrance, and deep, when the painful area is the cervix, bladder and/or the lower part of the pelvis.2 Another classification divides it into primary, associated with pain at the beginning of sexual life, and secondary, when it appears later.3 It directly affects physical health, as well as sexual and mental well-being. Consequently, it can lead to depression, anxiety and low self-esteem in women who experience it.4 Studies show an association between hyperactivity of the pelvic muscles and dyspareunia, which can have a significant impact on physical and mental health, leading to problems such as depression, anxiety, hypervigilance to pain, negative body image and low self-esteem, in addition to the possibility of leading to other sexual dysfunctions.5 Multidisciplinary treatment is highly recommended in this population and aims to address the various physical, emotional and behavioral aspects involved in sexual dysfunctions. This approach involves the collaboration of a team made up of specialized professionals, such as gynecologists, physiotherapists, sex therapists, psychologists and/or psychiatrists. Among these professionals, physiotherapy stands out as an intervention capable of improving sexual health, through individualized approaches for each patient. Considering that many patients with dyspareunia do not respond adequately to conventional drug therapy, there is a clear need to seek new therapeutic alternatives, such as photobiomodulation (PBM). Previous studies show positive results in the use of PBM in improving pain related to musculoskeletal and arthritic conditions. Furthermore, the application of PBM in the area of pelvic physiotherapy has been expanded. A study carried out by Lev-Sagie et al.6 showed positive results in the use of photobiomodulation in women with vestibulodynia, in relation to pain. Previous studies also indicate that intravaginal application of PBM has been effective in alleviating pain in conditions related to chronic pelvic pain, endometriosis, and pelvic pain of myofascial origin, which suggests that photobiomodulation may be a promising therapy for women with dyspareunia.7 ,8,9 In recent years, research has been carried out to investigate the presence and increase of inflammatory mediators in different painful musculoskeletal disorders10-14. A study that applied photobiomodulation to patients with low back pain observed changes in some biomarkers, in plasma or microdialysate, indicating that patients with low back pain who receive photobiomodulation may present changes in the levels of inflammatory mediators.15 But to date, few studies have been carried out on this topic, none of them applied to women with dyspareunia The scarcity of studies standardizing an application protocol, which observes time of effect and analysis of inflammatory biomarkers in the use of photobiomodulation in women with dyspareunia, justifies the need for research on the topic. Therefore, the objective of this study is to compare the effects of vulvar and intravaginal application of PBM compared to the sham group on the pain and sexual function of women with dyspareunia in the immediate post-intervention moments and in follow-ups of 15, 30, 90 and 180 days.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged between 18 and 45 years classified with dyspareunia criteria, according to the guidelines of the European Association of Urology guideline (2022)2, who report pain in relationship greater than 3 on the visual numeric pain scale at the beginning of participation in the research , who present sensitivity to unidigital palpation of the pelvic muscular wall (e.g., levator ani, coccygeus, obturator) and who report feeling pain during penetration for at least 6 months.

Exclusion Criteria:

* Women with a history of neurological or oncological diseases or bone fractures in the pelvic region, in addition to radiculopathies, decompensated heart disease or metabolic disorders, pregnant women, lactating women, women in menopause, women with difficulties in understanding written or spoken language, in use of photosensitizing drugs, who present an inflammatory condition or have used anti-inflammatories on the day of the evaluation, red flags (post-coital bleeding, abrupt unexplained weight loss, presence of a mass visible on ultrasound, macroscopic or microscopic hematuria), who have a diagnosis of painful bladder syndrome, irritable bowel syndrome, interstitial cystitis, fibromyalgia. Who have a history of spine surgery or have undergone any surgical intervention with general anesthesia in the last 120 days. Who is currently undergoing pelvic physiotherapy treatment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Visual numeric pain scale (VNS) | The visual pain scale will be evaluated at the beginning and at the end of each laser application, in addition to being applied immediately after the intervention and in follow-ups of 15, 30, 90 and 180 days.
  The number 0 represents no pain and, gradually, the increase in pain intensity is represented by the numerical increase on the scale (values from 1-3: mild pain; 4-6: moderate pain; and 7-10: severe pain). The primary outcome will be considered clinically significant if there is a reduction of at least 2 points in the overall severity of pain compared to baseline after 8 applications, in any of the time intervals measured.

SECONDARY OUTCOMES:
Female sexual function - IFSF | will be applied at six moments: before starting treatment, after the end of 8 treatment sessions and in follow-ups of 15, 30, 90 and 180 days.
  The Female Sexual Function Index (FSFI) is a brief questionnaire, which can be self-administered, and which aims to assess female sexual response in six domains: sexual desire, sexual arousal, vaginal lubrication, orgasm, sexual satisfaction and pain. To do this, it presents 19 questions that assess sexual function over the last four weeks. For each question there is an answer pattern whose options receive scores from 0 to 5 in an increasing manner in relation to the presence of the function questioned. Only in questions about pain the score is defined inverted. A total score is presented at the end of the application, resulting from the sum of the scores for each domain multiplied by a factor that homogenizes the influence of each domain on the total score.
Quality of life - SF-36 | will be applied at six moments: before starting treatment, after the end of 8 treatment sessions and in follow-ups of 15, 30, 90 and 180 days.
  It consists of a multidimensional questionnaire made up of 36 items, encompassed in 8 scales or domains, which are: functional capacity, physical aspects, pain, general health status, vitality, social aspects, emotional aspects and mental health. It presents a score that ranges from 0 (zero) to 100 (obtained through Raw Scale calculation), where zero corresponds to the worst general state of health and 100 corresponds to the best state of health.
Inflammatory markers - IL6, IL10 and prostaglandins | will be applied pre-intervention, after 4 interventions and at the end of 8 interventions
  To observe the inflammatory status of the volunteers, the plasma concentration of IL-6 and IL-10 will be measured using the ELISA immunoassay method according to the manufacturer's instructions.
  To observe the inflammatory status of the volunteers, the plasma concentration of PGE2 - Multi-Format ELISA Kit - K051-H1 / K051-H5 will be titrated by ELISA assays as indicated by the manufacturer
Satisfaction scale referred | It will be applied at the end of the 8 treatment sessions and in follow-ups of 15, 30, 90 and 180 days.
  A satisfaction scale referred to with the treatment will be applied where the volunteer will have to give a number from 1 to 10 to how satisfied she is with the result of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No